CLINICAL TRIAL: NCT04955639
Title: Pilot Randomized Controlled Trial of a Smart Phone-Based Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Marler, MD (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Marler, MD, Sr. Dir., Clinical and Medical Affairs, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C-650
Record Dates: First submitted 2021-06-17; First posted 2021-07-09 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant
Masking Description: Participant blinded to arm assignment but not to the smoking cessation program he/she is using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): A commercially available mobile phone app and program
  Interventions: Other: Control
- Pivot (Active Comparator): Pivot mobile phone app and program
  Interventions: Other: Pivot

INTERVENTIONS:
Other: Control — Standard of Care - Control Smoking Cessation Program
  Other Names: Standard of Care
  Arms: Control
Other: Pivot — Pivot Program Smoking Cessation Program
  Other Names: Pivot Program
  Arms: Pivot

SUMMARY:
Two-arm, parallel-group, non-crossover, single-center pilot randomized controlled trial, enrolling up to 180 participants to evaluate the effect of the Pivot smoking cessation program (intervention) compared to usual care (commercially available app smoking cessation program plus optional nicotine replacement therapy, control).

DETAILED DESCRIPTION:
The present pilot randomized controlled trial compares user engagement and retention, change in attitudes towards quitting smoking, change in smoking behavior and participant feedback in adult smokers randomized either to the Pivot (intervention) or commercially available (control) smoking cessation programs.

We aim to assess participants' use of Pivot program and commercially available program. There will be a focus on assessing use and engagement, changes in attitudes towards quitting smoking and changes in smoking behavior over the course of the 2-year study, as well as participant feedback on the set-up, design, use experience, and impact of each program.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years of age
* Current daily cigarette smokers (at least 5 cigarettes per day) for the past 12 months
* Plans to quit smoking in the next 30 days
* Resident of the United States
* Able to read and comprehend English
* Owns and uses a smart phone compatible with the study app (iPhone 5 and above with operating system (iOS) 12 and above, or, Android 7.0 and above with operating system Android 7.0 and above)
* Has daily internet access on smart phone
* Comfortable downloading and using smart phone apps
* Willing to sign the Informed Consent Form

Exclusion Criteria:

* Pregnancy (self-reported)
* Health contraindications to nicotine replacement therapy (NRT) use (irregular heartbeat, high blood pressure not controlled with medication, heart attack or stroke in last 2 months, pregnant or breast feeding, skin allergies to adhesive tape or serious skin problems, stomach ulcers, history of seizures)
* Using other smoking cessation support, including apps and/or actively taking medication to quit smoking
* Daily marijuana use
* Residence with another person who is a participant in this study
* Immediate family member is a participant in this study
* Failure to provide contact or collateral information, failure to verify email address, and/or failure to demonstrate videoconference capability
* Participation in a previous study sponsored by Carrot Inc.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marler, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Pivot Health Technologies, Inc., San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marler JD, Fujii CA, Utley MT, Balbierz DJ, Galanko JA, Utley DS. Long-Term Outcomes of a Comprehensive Mobile Smoking Cessation Program With Nicotine Replacement Therapy in Adult Smokers: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Sep 18;11:e48157. doi: 10.2196/48157. PMID 37585282
- [Derived] Marler JD, Fujii CA, Utley MT, Balbierz DJ, Galanko JA, Utley DS. Outcomes of a Comprehensive Mobile Smoking Cessation Program With Nicotine Replacement Therapy in Adult Smokers: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Nov 24;10(11):e41658. doi: 10.2196/41658. PMID 36257323

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Pivot
Started | 94 | 94
Completed Week 12 Survey | 91 | 92
Completed (n = 89 fully completed the week 26 questionnaire n = 1 partially completed the week 26 questionnaire) | 90 | 90
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Week 26 survey not completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Pivot | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (8.2) | 46.6 (10.1) | 46.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 104
  Male | 40 | 44 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 62 | 66 | 128
  Race/Ethnicity: Black | 21 | 15 | 36
  Race/Ethnicity: American Indian | 0 | 1 | 1
  Race/Ethnicity: Hispanic, Latino, or Spanish Origin | 5 | 8 | 13
  Race/Ethnicity: Asian | 1 | 0 | 1
  Race/Ethnicity: Native Hawaiian | 2 | 0 | 2
  Race/Ethnicity: Some other race | 1 | 2 | 3
  Race/Ethnicity: Prefer not to answer | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 94 | 94 | 188
Self-reported health [Count of Participants; unit: Participants]
  Excellent health | 1 | 4 | 5
  Very good health | 33 | 24 | 57
  Good health | 48 | 51 | 99
  Fair health | 12 | 14 | 26
  Poor health | 0 | 1 | 1
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 17.2 (8.5) | 18.0 (9.6) | 17.6 (9.0)
Years smoking [Mean (Standard Deviation); unit: years] | 25.8 (10.1) | 27.7 (10.4) | 26.8 (10.3)
Tobacco products used [Count of Participants; unit: Participants]
  Cigarettes only | 83 | 79 | 162
  Cigarettes + E-cigarettes/vaping | 5 | 10 | 15
  Cigarettes + Cigars | 2 | 1 | 3
  Cigarettes + E-cigarettes/vaping + Cigars | 1 | 1 | 2
  Cigarettes + Chew/snuff | 0 | 2 | 2
  Cigarettes + E-cigarettes/vaping + Chew/snuff | 1 | 0 | 1
  Cigarettes + E-cigarettes/vaping + Pipe | 1 | 0 | 1
  Cigarettes + Hookah + Cigars | 1 | 0 | 1
  Cigarettes + Hookah | 0 | 1 | 1
Difficulty to Quit (DTQ) [Mean (Standard Deviation); unit: score on a scale] — Difficulty to Quit (DTQ) = If you were to quit smoking right now, how difficult do you think it would be to stay smoke-free? (1 = Really hard to stay quit, 10 = Really easy to stay quit)
  score on a scale | 3.6 (2.6) | 3.5 (2.3) | 3.5 (2.5)
Success to Quit (STQ) [Mean (Standard Deviation); unit: score on a scale] — Success to Quit (STQ): If you were to quit smoking right now, how successful would you be? (1 = not at all successful; 10 = completely successful)
  score on a scale | 4.3 (2.3) | 4.6 (2.4) | 4.5 (2.4)
Smoking Abstinence Self-Efficacy Questionnaire (SASEQ) [Mean (Standard Deviation); unit: score on a scale] — Smoking Abstinence Self-Efficacy Questionnaire (SASEQ) is a 6-question questionnaire answered on a 5-point Likert scale (0-4) that results in a score from 0-24. A lower score represents lower self-efficacy in regards to quitting smoking, while a higher score represents greater self-efficacy in regards to quitting smoking.
  score on a scale | 11.5 (4.9) | 11.8 (4.7) | 11.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Average Total App Openings at 12 Weeks
Description: App/program engagement is assessed with the self-report of total app openings through the first 12 weeks of the program. Calculated by summing the number of weekly app openings reported by participants weekly.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: app openings
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
app openings | 86.5 (66.3) | 157.9 (210.6)

2. Secondary Outcome: Desire to Quit (Yes/no)
Description: desire to quit smoking, participant self-report, yes/no
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 88 | 91
Participants
  Participants who answered "yes" to having a desire to quit smoking | 88 | 91
  Participants who answered "no" to having a desire to quit smoking | 0 | 0

3. Secondary Outcome: Change in Expected Difficulty in Staying Quit
Description: Expected difficulty to stay quit from smoking. Participants asked: "How difficult do you think it would be to stay smoke free?". Participant self-report on scale 1-10 (1=Really hard to stay quit, 10=Really easy to stay quit)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
score on a scale
  Difficulty to quit 12 weeks | 5.2 (3.0) | 5.7 (3.1)
  Change in Difficulty to quit from baseline to 12 weeks | 1.7 (3.4) | 2.2 (3.7)

4. Secondary Outcome: Change in Confidence Levels Towards Quitting Smoking
Description: Expected success in quitting smoking. Asked: " If you were to quit smoking right now, how successful would you be?". Participant self-report, scale 1-10 (1=Not at all successful, 10=Completely successful).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
score on a scale
  Success to quit 12 weeks | 5.8 (3.1) | 6.6 (3.0)
  Change in Success to quit from baseline to 12 weeks | 1.6 (3.6) | 2.0 (3.6)

5. Secondary Outcome: Self-Reported Smoking Abstinence
Description: participant self-report of 7-day and 30-day point prevalence abstinence (PPA) from smoking cigarettes
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
Participants
  7-day PPA at 12 weeks | 26 | 33
  30-day PPA at 12 weeks | 21 | 27

6. Secondary Outcome: Self-Reported Smoking Abstinence
Description: participant self-report of 7-day and 30-day point prevalence abstinence (PPA) from smoking cigarettes
Time Frame: 26 weeks
Population: Number of participants analyzed is different due to Intention to Treat (ITT) vs. Responder analyses.
  ITT includes entire study population from the study arm, while responder only includes participants who completed the 26 week questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  7-day PPA at 26 weeks ITT | 25 | 34
  7-day PPA at 26 weeks Responder: number analyzed (Participants) | 90 | 90
  7-day PPA at 26 weeks Responder | 25 | 34
  30-day PPA at 26 weeks ITT | 21 | 30
  30-day PPA at 26 weeks Responder: number analyzed (Participants) | 90 | 90
  30-day PPA at 26 weeks Responder | 21 | 30

7. Secondary Outcome: Self-Reported Smoking Abstinence
Description: participant self-report of 7-day and 30-day point prevalence abstinence (PPA) from smoking cigarettes
Time Frame: 52 weeks
Population: Number of participants analyzed is different due to Intention to Treat (ITT) vs. Responder analyses.
  ITT includes entire study population from the study arm, while responder only includes participants who completed the 52 week questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  7-day PPA at 52 weeks ITT | 29 | 39
  7-day PPA at 52 weeks Responder: number analyzed (Participants) | 90 | 89
  7-day PPA at 52 weeks Responder | 29 | 39
  30-day PPA at 52 weeks ITT | 28 | 34
  30-day PPA at 52 weeks Responder: number analyzed (Participants) | 90 | 89
  30-day PPA at 52 weeks Responder | 28 | 34

8. Secondary Outcome: Self-Reported Abstinence From All Tobacco Products
Description: participant self report of no tobacco product use including: cigarettes, e-cigarettes/vaping, cigars, chew/snuff, pipe, and hookah
Time Frame: 12 weeks
Population: Number of participants analyzed is different due to Intention to Treat (ITT) vs. Responder analyses.
  ITT includes entire study population from the study arm, while responder only includes participants who completed the 12 week questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-report no tobacco use ITT | 25 | 31
  Self-report no tobacco use Responder: number analyzed (Participants) | 91 | 92
  Self-report no tobacco use Responder | 25 | 31

9. Secondary Outcome: Self-Reported Abstinence From All Tobacco Products
Description: as for outcome 8
Time Frame: 26 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-report no tobacco use ITT | 23 | 32
  Self-report no tobacco use Responder: number analyzed (Participants) | 90 | 90
  Self-report no tobacco use Responder | 23 | 32

10. Secondary Outcome: Self-Reported Abstinence From All Tobacco Products
Description: as for outcome 8
Time Frame: 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-report no tobacco use ITT | 27 | 33
  Self-report no tobacco use Responder: number analyzed (Participants) | 90 | 89
  Self-report no tobacco use Responder | 27 | 33

11. Secondary Outcome: Biochemically Confirmed Abstinence
Description: Participants who report they have achieved at least 7-day point prevalence abstinence at 12 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Time Frame: 12 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Biovalidated abstinence ITT | 12 | 27
  Biovalidated abstinence Responder: number analyzed (Participants) | 91 | 92
  Biovalidated abstinence Responder | 12 | 27

12. Secondary Outcome: Biochemically Confirmed Abstinence
Description: Participants who report they have achieved at least 7-day point prevalence abstinence at 26 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Time Frame: 26 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Biovalidated abstinence ITT | 14 | 26
  Biovalidated abstinence Responder: number analyzed (Participants) | 90 | 90
  Biovalidated abstinence Responder | 14 | 26

13. Secondary Outcome: Biochemically Confirmed Abstinence
Description: Participants who report they have achieved at least 7-day point prevalence abstinence at 52 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Time Frame: 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Biovalidated abstinence ITT | 17 | 29
  Biovalidated abstinence Responder: number analyzed (Participants) | 90 | 89
  Biovalidated abstinence Responder | 17 | 29

14. Secondary Outcome: Self-Reported Continuous Abstinence
Description: Defined as self-report of 7-day PPA or greater at 12 weeks, 30-day PPA at 26 weeks, and no more than 5 cigarettes during the intervening time period.
Time Frame: 26 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-reported continuous abstinence ITT | 15 | 24
  Self-reported continuous abstinence Responder: number analyzed (Participants) | 90 | 90
  Self-reported continuous abstinence Responder | 15 | 24

15. Secondary Outcome: Self-Reported Continuous Abstinence
Description: as for outcome 14
Time Frame: 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-reported continuous abstinence ITT | 8 | 19
  Self-reported continuous abstinence Responder: number analyzed (Participants) | 90 | 89
  Self-reported continuous abstinence Responder | 8 | 19

16. Secondary Outcome: Biochemically Confirmed Continuous Abstinence
Description: Defined as self-report of smoking no more than five cigarettes from 12 weeks after enrollment, and biochemical confirmation of abstinence on all previous and present biovalidation tests, with biochemical confirmation defined as:
  Participants who report they have achieved at least 7-day point prevalence abstinence at 12 weeks and 26 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Time Frame: 26 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Biochemically confirmed continuous abstinence ITT | 9 | 20
  Biochemically confirmed continuous abstinence Responder: number analyzed (Participants) | 90 | 90
  Biochemically confirmed continuous abstinence Responder | 9 | 20

17. Secondary Outcome: Biochemically Confirmed Continuous Abstinence
Description: Defined as self-report of smoking no more than five cigarettes from 12 weeks after enrollment, and biochemical confirmation of abstinence on all previous and present biovalidation tests, with biochemical confirmation defined as:
  Participants who report they have achieved at least 7-day point prevalence abstinence at 12 weeks, 26 weeks, and 52 weeks will undergo a videoconference visit with study staff in which they provide a witnessed breath sample using a provided personal mobile carbon monoxide breath sensor. Breath sample values less than 10 ppm (parts per million) will be considered consistent with biochemical abstinence.
Time Frame: 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Biochemically confirmed continuous abstinence ITT | 8 | 18
  Biochemically confirmed continuous abstinence Responder: number analyzed (Participants) | 90 | 89
  Biochemically confirmed continuous abstinence Responder | 8 | 18

18. Secondary Outcome: Proportion With ≥ 50% CPD Reduction
Description: The proportion of participants who reduced their cigarettes per day (CPD) by ≥ 50% compared to baseline
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 90 | 90
Participants | 59 | 56

19. Secondary Outcome: User Satisfaction - User Feedback
Description: User satisfaction with the smoking cessation program, specifically its impact on motivation to quit smoking, and the amount of cigarettes smoked per day. Participants were asked: "How has using your assigned program affected your motivation to quit smoking?" and "How has using your assigned program affected the number of cigarettes you smoke per day?" with the answer choices of "increased", "not affected", and "decreased".
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 92 | 92
Participants
  How has using your assigned program affected your motivation to quit smoking?: increased | 54 | 72
  How has using your assigned program affected your motivation to quit smoking?: not affected | 35 | 19
  How has using your assigned program affected your motivation to quit smoking?: decreased | 3 | 1
  How has using your assigned program affected the number of cigarettes you smoke per day?: increased | 2 | 2
  How has using your assigned program affected the number of cigarettes you smoke per day?: not affected | 34 | 25
  How has using your assigned program affected the number of cigarettes you smoke per day?: decreased | 56 | 65

20. Secondary Outcome: Additional User Feedback
Description: User feedback on what they have learned from using their assigned smoking cessation program. Participants were asked "Which of the following best described what you have learned from using your program?" with the answer choices: "I've learned some really unique/key insights into my smoking behavior", "I've learned some things but nothing that impactful", "I have not learned anything from the program", and "I am more confused after using the program".
Time Frame: 3 weeks
Population: Participants that completed the 3 week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 90 | 89
Participants
  I've learned some really unique/key insights into my smoking behavior | 51 | 72
  I've learned some things but nothing that impactful | 26 | 16
  I have not learned anything from the program | 12 | 1
  I am more confused after using the program | 1 | 0

21. Secondary Outcome: User Feedback - Setup and Starting the Program
Description: User feedback with the smoking cessation program, specifically ease of set-up and starting of the program (scale of 1-10, higher value equates to easier time setting up and starting use of the program)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
score on a scale | 7.1 (3.0) | 8.2 (2.3)

22. Secondary Outcome: User Feedback
Description: User feedback with the smoking cessation program, specifically whether the program helped with their smoking cessation goals (true/false), and whether the program helped them quit smoking (true/false).
Time Frame: 26 weeks
Population: Number of participants differs per question:
  Only participants reporting 7-day PPA (n=25 control, n=34 Pivot) were asked if their study program helped them quit smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
Participants
  Study program helped them with their goals related to smoking - answered "true" | 69 | 79
  Among participants reporting 7-day PPA: study program helped them quit smoking - answered "true": number analyzed (Participants) | 25 | 34
  Among participants reporting 7-day PPA: study program helped them quit smoking - answered "true" | 22 | 34

23. Secondary Outcome: User Feedback: Number of Participants Who Agreed That Their Program Helped Them Quit Smoking
Description: User feedback with the smoking cessation program, specifically whether the program helped them quit smoking (true/false).
Time Frame: 52 weeks
Population: Only participants reporting 7-day PPA at 52 weeks (n=29 control, n=39 Pivot) were asked if their study program helped them quit smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 29 | 39
Participants | 26 | 35

24. Secondary Outcome: User Satisfaction - Net Promoter Score (NPS)
Description: User satisfaction with the smoking cessation program, specifically the likelihood of recommending the program to a friend. Measured with a net promoter score (NPS).
  Participants are asked "How likely are you to recommend your study program to a friend or colleague?" and answer on a 10-point (1-10) scale (where 1=Not at all likely and 10=Very likely).
  NPS was calculated for each study group by subtracting the percentage of respondents who answered ≤6 (detractors) from the percentage of respondents who answered 9 or 10 (promotors).
  NPS formula = %promotor - %detractor NPS has a score range between -100 and 100 (-100 indicates 100% detractors, 100 indicated 100% promotors of the program).
  A higher NPS score indicates greater promoters of the program, and thus a greater likelihood of individuals recommending the program to a friend.
Time Frame: 4 weeks, 12 weeks, and 26 weeks
Population: Number analyzed differs based on differential completion of the surveys at each of the timepoints: 4 weeks, 12 weeks, and 26 weeks
Measure: Number; unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
score on a scale
  NPS score at 4 weeks: number analyzed (Participants) | 88 | 91
  NPS score at 4 weeks | 1.1 | 50.6
  NPS score at 12 weeks | 11.0 | 44.6
  NPS score at 26 weeks: number analyzed (Participants) | 89 | 90
  NPS score at 26 weeks | 23.6 | 57.8

25. Secondary Outcome: Engagement With Program - Number of Times App Was Opened
Description: Collected weekly during the first 12 weeks after enrollment:
  o Number of times app opened
  Average number of times the app was opened, cumulative over 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: number of app openings
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
number of app openings | 86.5 (66.3) | 157.9 (210.6)

26. Secondary Outcome: Engagement With Program - Number of Days App Was Opened
Description: Collected weekly during the first 12 weeks after enrollment:
  o Number of days in which app was opened
  Average number of days the app was opened, cumulative over 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
days | 50.4 (25.2) | 49.6 (24.1)

27. Secondary Outcome: Engagement With Program - Number of Weeks App Was Opened
Description: Collected weekly during the first 12 weeks after enrollment:
  o Number of weeks in which app was opened
  Average number of weeks the app was opened, cumulative over 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
weeks | 11.0 (2.3) | 11.0 (2.2)

28. Secondary Outcome: Participant Changes in Self-Efficacy
Description: 6-item Smoking Abstinence Self-efficacy Questionnaire (SASEQ) (Spek V, et al. Int.J. Behav. Med. (2013) 20:444-449).
  SASEQ score is on a scale of 0-24. Each of the 6 questions is answered on a 5-point Likert scale (0-4). Greater scores indicate greater self-efficacy toward quitting smoking.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 91 | 92
score on a scale
  SASEQ 12 weeks | 14.1 (6.2) | 14.5 (6.9)
  Change in SASEQ from baseline to 12 weeks | 2.7 (7.9) | 2.6 (6.7)

29. Secondary Outcome: Participant Changes in Self-Efficacy
Description: as for outcome 28
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Pivot
Number analyzed (Participants) | 90 | 89
score on a scale
  SASEQ 52 weeks | 12.6 (8.1) | 14.9 (7.9)
  Change in SASEQ from baseline to 52 weeks | 1.0 (8.5) | 3.2 (7.8)

30. Secondary Outcome: Participant Changes in Self-reported Health and Wellbeing
Description: participant self-report, choices for reporting health: excellent, very good, good, fair, or poor
Time Frame: 12 weeks
Population: Participant numbers are different from baseline to week 26 due to 4 participants from each arm not completing the week 16 questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Self-reported health at baseline: Excellent | 1 | 4
  Self-reported health at baseline: Very good | 33 | 24
  Self-reported health at baseline: Good | 48 | 51
  Self-reported health at baseline: Fair | 12 | 14
  Self-reported health at baseline: Poor | 0 | 1
  Self-reported health at 12 weeks: number analyzed (Participants) | 90 | 90
  Self-reported health at 12 weeks: Excellent | 6 | 4
  Self-reported health at 12 weeks: Very good | 27 | 25
  Self-reported health at 12 weeks: Good | 37 | 42
  Self-reported health at 12 weeks: Fair | 18 | 18
  Self-reported health at 12 weeks: Poor | 2 | 1

31. Secondary Outcome: Self-Reported Nicotine Replacement Therapy (NRT) Use
Description: Nicotine replacement therapy (NRT) use assessed with participant orders of NRT
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  ≥1 NRT single-therapy order | 8 | 23
  ≥1 NRT combination-therapy order | 57 | 44
  ≥1 NRT single-therapy order + ≥1 NRT combination-therapy order | 12 | 26
  No orders | 17 | 1

32. Secondary Outcome: Self-Reported Nicotine Replacement Therapy (NRT) Use
Description: Nicotine replacement therapy (NRT) use assessed with participant orders of NRT
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  ≥1 NRT single therapy order | 9 | 22
  ≥1 NRT combination therapy order | 57 | 42
  ≥1 NRT single therapy + ≥1 NRT combination therapy order | 14 | 29
  None | 14 | 1

33. Secondary Outcome: Adverse Events
Description: participant self-report of adverse events and any issues experienced with assigned study app/program as well as the provided nicotine replacement therapy (NRT). For further adverse event details - see adverse event portion of this record.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Pivot
Number analyzed (Participants) | 94 | 94
Participants
  Participants who experienced adverse events/issues with their assigned study program | 0 | 0
  Participants who experienced adverse events/issues with nicotine replacement therapy | 17 | 19

ADVERSE EVENTS:
Time Frame: Participants self-report adverse event experienced due to their assigned program and/or the NRT that they ordered during the study. Participants were asked at 12 weeks and 26 weeks if they had any issues with their assigned program and/or with their use of nicotine replacement therapy.
Arm/Group | Control | Pivot
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/94
Other Adverse Events (participants affected / at risk) | 17/94 | 19/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=94) | Pivot (N=94)
GI upset due to NRT lozenge or gum use (Gastrointestinal disorders) | 1 (1) | 6 (6)
Skin irritation due to NRT patch use (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)
Heartburn due to NRT lozenge or gum use (Gastrointestinal disorders) | 3 (3) | 0 (0)
Sleep issues - wild dreams, insomnia (General disorders) | 3 (3) | 3 (3)
Headache due to NRT use (General disorders) | 1 (1) | 1 (1)
Hiccups due to NRT lozenge or gum use (Gastrointestinal disorders) | 0 (0) | 2 (2)
Jittery, racing heart, or lightheaded feeling due to NRT use (General disorders) | 1 (1) | 2 (2)
Mouth irritation or sore throat due to NRT lozenge or gum use (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT04955639/Prot_SAP_001.pdf